CLINICAL TRIAL: NCT02950116
Title: Lung Clearance Index in Pediatric Patients With Obstructive Lung Disease
Brief Title: Lung Clearance Index (LCI) in Pediatric Patients With Obstructive Lung Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Availabe time for inclusion ended (master thesis)
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LCI-OLD-ped
Record Dates: First submitted 2016-10-11; First posted 2016-10-31 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-05

CONDITIONS: Asthma; Bronchiectasis; Cystic Fibrosis
MeSH Terms: conditions — Asthma; Bronchiectasis; Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Asthma (Active Comparator): Asthmatic patients will perform three multiple breath nitrogen washout tests (N2-MBW-test)
  Interventions: Device: Perform three multiple breath nitrogen washout tests (N2-MBW-test)
- Non-CF bronchiectasis (Active Comparator): Patients with non-CF bronchiectasis will perform three multiple breath nitrogen washout tests (N2-MBW-test)
  Interventions: Device: Perform three multiple breath nitrogen washout tests (N2-MBW-test)
- Cystic fibrosis (Active Comparator): Patients with cystic fibrosis will perform three multiple breath nitrogen washout tests (N2-MBW-test)
  Interventions: Device: Perform three multiple breath nitrogen washout tests (N2-MBW-test)

INTERVENTIONS:
Device: Perform three multiple breath nitrogen washout tests (N2-MBW-test) — * Patient is sitting in upright position, nose clip in place and breathing through a mouth piece with filter (neither sitting forward with back bent, nor supporting arms such that shoulders are raised)
  * Patient's breathing pattern is stable for a minimum of 5 breaths
  * Start of washout by inhaling 100% oxygen (initiated by lab technician)
  * Continuous stable breathing pattern until end of washout test
  * End target = 1/40th of start N2 concentration
  * To ensure end of washout is achieved, patients should breathe 5 more breaths below the target concentration before the trial is terminated
  * Three N2-MBW-tests are performed consecutively. Time between each test is [duration of the previous test*1.5] (e.g. test duration = 6 min., time to next test = 6*1.5 = 9 min.)

SUMMARY:
Chronic respiratory diseases (CRDs) affect the airways and other structures of the lungs and thereby lead to ventilation inhomogeneity. The most common CRDs in children are asthma, bronchiectasis and cystic fibrosis (CF). All three are obstructive diseases. However, while asthma is mostly characterized by obstruction due to bronchoconstriction of the airways, obstruction in bronchiectasis and CF originates primarily from mucus retention due to abnormal airway clearance mechanisms.

The Nitrogen Multiple Breath Washout test (N2-MBW-test) is a robust and sensitive detector of early pulmonary changes and ventilation inhomogeneity. The minimal cooperation which is required for this test makes it very convenient for use in any age category.

Research on LCI described it as a reliable indicator of obstructive lung disease in pediatric CF patients as from 6 years of age. Whether LCI is a reliable parameter for early lung disease in asthma children is less clearly demonstrated. No data were found on LCI calculated from the N2-MBW-test in children with bronchiectasis.

DETAILED DESCRIPTION:
Subjects of all the intervention groups will perform three consecutive nitrogen multiple breath washout tests (N2-MBW-tests) when attending the Universitair Ziekenhuis Brussel (UZB) for their scheduled pulmonology consultation. Only the best measurement (based on LCI result) will be taken into account when comparing the groups. Every subject will be positioned in the same seated position.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable asthma
* Patients with non-CF bronchiectasis
* Patients with cystic fibrosis
* Aged 6-17 years
* FEV1 (%pred) >50%
* Written informed consent from the parents or legal guardian

Exclusion Criteria:

* Unstable disease (e.g. pulmonary exacerbation, acute deterioration, acute asthma crisis)
* Patients mentally not capable to participate in the study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-04-07 (Actual)

PRIMARY OUTCOMES:
LCI | Day 1
  LCI will be calculated from the 3 N2-MBW-tests. The test with the lowest LCI will be used for analysis of the other outcome measurements.

SECONDARY OUTCOMES:
S_cond | Day 1
  S_cond will be calculated from the N2-MBW-test with the lowest LCI
S_acin | Day 1
  S_acin will be calculated from the N2-MBW-test with the lowest LCI
Duration of the N2-MBW-test | Day 1
  Duration of the N2-MBW-test with the lowest LCI will be taken into account for analysis
Number of washout breaths | Day 1
  Will be determined at the end of the N2-MBW-test
FRC | Day 1
  FRC will be calculated from the N2-MBW-test

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke Eyns, MSc, PT, Principal Investigator — UZ Brussel Laarbeeklaan 101 1090 Brussels Belgium
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No